CLINICAL TRIAL: NCT05592808
Title: Comparison of the Effects of Low-Dye and Kinesio Taping Methods in Plantar Fasciitis
Brief Title: Comparison of Taping Techniques in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KaratayESWT
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-10

CONDITIONS: Plantar Fasciitis; Pain; Foot Diseases
MeSH Terms: conditions — Fasciitis, Plantar; Pain; Foot Diseases | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dye Taping (Experimental): In addition to the ESWT applied to the participants in the control group, Low-Dye Taping will be applied to the participants in this group once a week for 3 sessions.
  Interventions: Device: Extracorporeal Shockwave Therapy (ESWT); Other: Low-Dye Taping
- Kinesio Taping (Experimental): In addition to the ESWT applied to the participants in the control group, Kinesio Taping will be applied to the participants in this group once a week for 3 sessions.
  Interventions: Device: Extracorporeal Shockwave Therapy (ESWT); Other: Kinesio Taping
- Extracorporeal Shockwave Therapy (ESWT) (Active Comparator): Participants in the control group will receive 3 sessions of ESWT once a week.
  Interventions: Device: Extracorporeal Shockwave Therapy (ESWT)

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy (ESWT) — Extracoporeal shock wave, 2000 shots/time, once a week for 3 weeks, shock wave freqency: 10Hz, total energy: 166 mJ/mm2, Pressure 2.5 Bar
Other: Low-Dye Taping — After ESWT application, Low-Dye Taping will be applied 3 times, once a week.
  Arms: Low-Dye Taping
Other: Kinesio Taping — After ESWT application, Kinesio Taping will be applied 3 times, once a week.
  Arms: Kinesio Taping

SUMMARY:
The aim of this study is to investigate the effects of Low-Dye and Kinesio Taping on pain and function in individuals with plantar fasciitis.

DETAILED DESCRIPTION:
Subject: In this study, the effects of Low-Dye Taping and Kinesio Taping (KT) on pain and function will be investigated in individuals with plantar fasciitis. There are studies on both Low-Dye banding and KT in the literature and they are popular applications recently. However, to the best of our knowledge, when we look at the Turkish and English literature, no study has been found comparing these two therapeutic massages in terms of pain, functionality and performance.

Purpose: Plantar fasciitis (PF) is a clinical picture characterized by degeneration of the plantar fascia resulting from repetitive microtrauma to the plantar fascia causing an inflammatory reaction. It is one of the most common causes of heel pain in adults. The plantar fascia has a fundamental role in the biomechanics of the foot, supporting the medial longitudinal arch (MLA), distributing forces and stresses of the foot during gait or other loading conditions. Disorders in the musculoskeletal and somatosensory system in patients with plantar fasciitis may cause pain and decrease in functional capacity. Therefore, its purpose is; This study was planned to show the effectiveness of taping methods applied in addition to ESWT in individuals presenting with heel pain. Thanks to the findings to be obtained from our study, it is aimed to contribute to the literature with objective, evidence-based results in this field.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with plantar fasciitis by a physician
* Age between 18 and 30 years
* Agree to participate in the study

Exclusion Criteria:

* Not having surgery
* Disagree to participate in the study
* Infection
* Pregnancy
* Tumor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain at 3 Session | Changes in the VAS scores of the three groups before the treatment
  A visual analog scale (VAS) numbered 0-10 will be used in the assessment of pain.
Change from baseline in Pain at 3 Session | Changes in the AOFAS scores of the three groups before the treatment
  In functional evaluation, the scale developed by The American Orthopaedic Foot & Ankle Society (AOFAS) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Sönmez ÜNÜVAR, Principal Investigator — KTO Karatay University
Locations (2):
- Turkey (Türkiye) (2):
  - KTO Karatay University, Konya
  - Bayram Sönmez ÜNÜVAR, Konya

IPD SHARING:
Plan to Share IPD: No